CLINICAL TRIAL: NCT04093869
Title: Improving Lung Transplant Outcomes With Coping Skills and Physical Activity
Acronym: INSPIRE-III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00100300
Record Dates: First submitted 2019-09-06; First posted 2019-09-18 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Post-Lung Transplantation
MeSH Terms: interventions — Exercise; Standard of Care; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping Skills Training combined with Exercise (CSTEX) (Experimental): The CSTEX intervention will consist of 12, 30 minute weekly sessions conducted by a respiratory therapist knowledgeable about lung transplantation and trained in motivational interviewing, Cognitive Behavioral Therapy (CBT), and exercise therapy.
  Interventions: Behavioral: Coping Skills Training combined with Exercise (CSTEX)
- Standard of Care plus Education (SOC-ED) (Experimental): The SOC-ED intervention will consist of 12, 30 minute weekly sessions conducted by a health educator knowledgeable about transplantation and skilled in educational instruction.
  Interventions: Behavioral: Standard of Care plus Education (SOC-ED)

INTERVENTIONS:
Behavioral: Coping Skills Training combined with Exercise (CSTEX) — The CSTEX condition has two integrated components: the CST component will systematically train patients in the use of coping skills for stress reduction and promote key transplant-specific health behaviors. The exercise component of the intervention will progressively increase participants exercise and promote daily physical activity through motivational interviewing strategies.
  Arms: Coping Skills Training combined with Exercise (CSTEX)
Behavioral: Standard of Care plus Education (SOC-ED) — The SOC-ED condition provides support and enhanced post-transplant education. Participants will be given detailed educational information about post-transplant care, the importance of medication adherence, and maintenance of physical activity.
  Arms: Standard of Care plus Education (SOC-ED)

SUMMARY:
This study evaluates the effectiveness of a coping skills and exercise (CSTEX) intervention among post lung transplant patients aimed to reduce distress and improve functional capacity. Half of the patients will receive CSTEX and half will receive the standard of care plus transplant education (SOC-ED).

DETAILED DESCRIPTION:
The study will aim to evaluate the effectiveness of the CSTEX intervention in (i) reducing distress and (ii) improving functional capacity. It is hypothesized that compared to SOC-ED, the CSTEX intervention will result in 1) greater reductions in global distress measured by an established psychometric test battery; and 2) greater improvements in functional capacity assessed by distance walked on a standard Six Minute Walk test (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* Single or bilateral first lung transplant recipient; discharged from the hospital and at least 6 weeks post-transplant; completed post-transplant pulmonary rehabilitation within the past 18 months; on stable medication regimen; proficient in the English language

Exclusion Criteria:

* Illness such as malignancies that are associated with a life-expectancy of < 12 months; current pregnancy; inability to read or to provide informed consent; multi-organ transplant recipient or repeat lung transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blumenthal JA, Mabe S, Arthur D, Frankel C, McKee DC, Morrison S, Sherwood A, Snyder LD, Palmer SM; INSPIRE III Investigators. Telehealth interventions to improve outcomes in lung transplant recipients: Primary results of the INSPIRE-III randomized clinical trial. J Heart Lung Transplant. 2025 Sep;44(9):1449-1459. doi: 10.1016/j.healun.2025.03.017. Epub 2025 Apr 1. PMID 40180232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned in a 1:1 ratio to either CSTEX condition delivered over the telephone or to a standard of care plus transplant education (SoC-ED) control condition.
Period: Overall Study
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Started | 90 | 90
Completed | 89 | 89
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED) | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 60 (12) | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 55 | 53 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 89 | 88 | 177
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 14 | 25
  White | 77 | 74 | 151
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Psychological Distress
Description: A composite distress score will assess change from baseline to 12 weeks (post-intervention) and combine the following instruments: General Health Questionnaire, Perceived Stress Scale, Beck Depression Inventory-II, State Trait Anxiety Inventory, and PROMIS Anger. The composite distress score is the average of the participant's rank for change (from baseline to 12 weeks) on each of the 5 scales. A lower rank represents more improvement (decrease in global distress) and higher ranks represent less improvement (or worsening of distress). Scoring is based on the number of participants analyzed; in this case the possible score range is 1-180. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: 3 participants were excluded because they had missing values for at least one of the instruments that contributed to the composite distress score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 88 | 89
units on a scale | 91 (40) | 87 (33)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; p = 0.40, Regression, Linear — Not adjusted for multiple comparisons. Full alpha of 0.05 was allocated to this as the sole primary outcome; Mean Difference (Net) = 4.1, 95% CI 2-sided [-6 to 14], Standard Error of Mean 5.1 — A negative mean difference would represent a better outcome in the CSTEX arm compared to the SOC-ED arm

2. Secondary Outcome: Change in Functional Capacity
Description: Functional capacity will be measured by distance walked on a standard Six Minute Walk Test (6MWT) at baseline and again post-intervention at 12 weeks. Distance measured in feet. Greater distance represents better functional capacity. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: Assessment of functional capacity was limited due to the inability of participants to attend in person visits during COVID-19. Seventy-one participants were unable to complete the 6MWT at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 52 | 57
feet | 1451 (332) | 1472 (262)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = 20.7, 95% CI 2-sided [-44 to 85], Standard Error of Mean 32.6 — A positive value for the estimate represents a greater distance walked for the CSTEX arm compared to the SOC-ED arm

3. Secondary Outcome: Change in Physical Activity
Description: Daily physical activity (average steps per day) will be assessed via a wrist-worn activity monitor (Actigraph GT9X Link) for 7 consecutive days at baseline and again post-intervention at 12 weeks. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: 5 participants had missing data for the baseline and/or post-intervention physical activity (steps) measurement.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 87 | 88
steps per day | 8037 (3103) | 8612 (3161)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Median Difference (Net) = -316, 95% CI 2-sided [-979 to 346], Standard Error of Mean 336 — A positive value for the estimate would represent more steps per day for the CSTEX arm compared to the SOC-ED arm

4. Secondary Outcome: Change in Sleep Quality
Description: Sleep quality (average total minutes of sleep per night) will be assessed via the Pittsburgh Sleep Quality Index at baseline and again post-intervention at 12 weeks. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: 8 participants were missing a PSQI score at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 86 | 86
minutes per night | 421 (92) | 401 (66)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = 14.7, 95% CI 2-sided [-5 to 34], Standard Error of Mean 10

5. Secondary Outcome: Change in Quality of Life
Description: Quality of Life will be assessed via the Lung Transplant Quality of Life Survey, which is comprised of 10 scales that measure symptoms, health perceptions, functioning, and well being at baseline and again post-intervention at 12 weeks. The QOL overall score ranges from 1 to 5, with a higher score indicating worse health. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: Two participants were missing a QOL score at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 89 | 89
score on a scale | 1.78 (0.49) | 1.78 (0.56)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = 0.0034, 95% CI 2-sided [-0.1 to 0.11], Standard Error of Mean 0.055 — A negative value for the estimate would represent a better QOL survey score for the CSTEX arm compared to the SOC-ED arm

6. Secondary Outcome: Change in Frailty
Description: Frailty will be measured by performance on the Fried Frailty Index. This assessment includes measures on patient's weight, exhaustion level, physical activity, walking speed, and hand grip strength at baseline and again post-intervention at 12 weeks. Scores range from 0 to 5, with lower scores indicating less frailty. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: Assessment of frailty was limited due to the inability of participants to attend in person visits during COVID-19. Sixty-eight participants were missing the Fried Frailty Index measurement at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 54 | 58
score on a scale | 0.62 (0.74) | 0.52 (0.73)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = 0.041, 95% CI 2-sided [-0.22 to 0.30], Standard Error of Mean 0.13 — A negative value for the estimate would represent a better Frailty index score for the CSTEX arm compared to the SOC-ED arm

7. Secondary Outcome: Change in Problem-Focused Coping
Description: Coping was assessed via the Brief COPE Inventory, which is composed of scales that measure problem-focused coping, emotion-focused coping, and avoidant coping responses at baseline and again post-intervention at 12 weeks. Items are scored on a 4-point Likert scale, with 1 indicating a coping mechanism that the participant has not been doing at all, to 4 indicating a coping mechanism in which the participant has been doing a lot. A higher average score within the problem-focused subscale indicates better coping strategies. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: Two participants were missing a Brief COPE score at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 89 | 89
score on a scale | 2.64 (0.79) | 2.73 (0.79)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.20 to 0.17], Standard Error of Mean 0.09

8. Secondary Outcome: Change in Emotion-Focused Coping
Description: Coping was assessed via the Brief COPE Inventory, which is composed of scales that measure problem-focused coping, emotion-focused coping, and avoidant coping responses at baseline and again post-intervention at 12 weeks. Items are scored on a 4-point Likert scale, with 1 indicating a coping mechanism that the participant has not been doing at all, to 4 indicating a coping mechanism in which the participant has been doing a lot. A higher score within the emotion-focused coping subscale indicates better coping strategies. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: Two participants were missing a Brief COPE score at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 89 | 89
score on a scale | 2.26 (0.51) | 2.25 (0.49)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.13 to 0.10], Standard Error of Mean 0.06

9. Secondary Outcome: Change in Avoidant Coping
Description: Coping was assessed via the Brief COPE Inventory, which is composed of scales that measure problem-focused coping, emotion-focused coping, and avoidant coping responses at baseline and again post-intervention at 12 weeks. Items are scored on a 4-point Likert scale, with 1 indicating a coping mechanism that the participant has not been doing at all, to 4 indicating a coping mechanism in which the participant has been doing a lot. A lower score within the avoidant coping subscale indicates a more useful coping strategy. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: Two participants were missing a Brief COPE score at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 89 | 89
score on a scale | 1.45 (0.36) | 1.46 (0.34)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.12 to 0.07], Standard Error of Mean 0.05

10. Secondary Outcome: Change in Self-Efficacy
Description: Self-efficacy will be assessed via the General Self-Efficacy Scale, which is a 10-item scale that measures emotional distress at baseline and again post-intervention at 12 weeks. Scores range from 10-40 with a higher score indicating better self-efficacy. The change value is calculated as T2 (12 weeks) - T1 (baseline).
Time Frame: Baseline to 12 weeks
Population: 5 participants were missing a GSE score at baseline and/or post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
Number analyzed (Participants) | 89 | 86
score on a scale | 33.3 (5.1) | 33.1 (4.7)
Statistical Analysis 1: Comparison: Coping Skills Training Combined With Exercise (CSTEX) vs Standard of Care Plus Education (SOC-ED); Test type: Superiority; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.83 to 1.60], Standard Error of Mean 0.62 — A positive value for the estimate represents better self-efficacy for the CSTEX arm compared to the SOC-ED arm

11. Secondary Outcome: Chronic Lung Allograft Dysfunction (CLAD) Free Survival
Time Frame: Up to 3 years post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through post-intervention assessments, approximately 12 weeks
Description: The only Adverse Events collected were hospitalization and death.
Arm/Group | Coping Skills Training Combined With Exercise (CSTEX) | Standard of Care Plus Education (SOC-ED)
All-Cause Mortality (participants affected / at risk) | 0/90 | 1/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04093869/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04093869/ICF_000.pdf